CLINICAL TRIAL: NCT00987025
Title: Technologies for Enhancing Access and Health Management
Brief Title: Initial Evaluation of Telehealth Blood Pressure Stations in Nutrition Centers
Acronym: TEAhM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LeadingAge (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Wright State University (Other); Healthanywhere Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HHSA290200600024I, TO #2; HHSA29032001T
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: hypertension; telehealth; nurse monitor; nutrition center
MeSH Terms: conditions — Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telehealth (Experimental): Telehealth participants will be recruited from centers that have a telehealth blood pressure station installed. Participants will be asked to use the station once per week. Blood pressure measures will be monitored by nurse researchers - out of range values will result in appropriate medical recommendations.
  Interventions: Behavioral: Telehealth
- Control (Active Comparator): Control participants will receive education material.
  Interventions: Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Telehealth — Use of telehealth blood pressure station every week
  Arms: Telehealth
Behavioral: Educational materials — Control
  Arms: Control

SUMMARY:
The purpose of TEAhM is to determine if telehealth blood pressure stations can be installed and used in senior nutrition centers and to do a preliminary comparison of blood pressure outcomes among nutrition center clients who use the telehealth blood pressure stations compared to participants who do not use the stations. Specifically, the goals of the project are to determine if these monitors can be successfully implemented in this community-based setting, the degree to which older adults with hypertension are comfortable using the technology, and whether remote nurse monitoring of blood pressure using this technology is a feasible supplement to office-based care.

DETAILED DESCRIPTION:
TEAhM will be conducted in four senior nutrition centers in the state of Ohio. Using these facilities as field centers, we will recruit 144 older, hypertensive adults who receive nutrition assistance at these centers. Wright State staff will obtain permission from enrolled participants in the intervention centers to contact primary care physicians for the purpose of obtaining recommended intervention protocols and defining referral criteria for changes in blood pressure treatment. We will install telehealth kiosks at two of the four nutrition centers. Participants who enroll at the two centers with kiosks will be considered "intervention participants" and those who enroll at the two centers without the kiosks will be considered "control participants." The kiosks will enable participants to conduct self-monitoring of their blood pressure at the nutrition facility. Blood pressure data from intervention participants will be sent to a central server managed by Healthanywhere, the telehealth partner in this project. Nurse-researchers from WSU will receive email alerts about out of range blood pressure measures, monitor blood pressure readings once a week, and make referrals for medical care according to criteria defined by participants' primary care physicians at the time of enrollment. Control and intervention participants will receive educational materials on general wellness that are publicly available.

Demographic information, background health, comfort with technology, and baseline blood pressure measures will be collected at baseline in on paper forms by WSU nurse researchers. Follow up blood pressure measures and other health utilization measures and reported health events will be collected from both intervention and control facilities during follow-up phone contacts with study personnel every two months. Blood pressure will be measured for all participants at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55 years
* Current use of nutrition center resources ≥1 time/week
* Physician-diagnosed hypertension
* Clinically stable if on oral therapy
* Physician willingness to interact with nurse reviewers (intervention arm only)

Exclusion Criteria:

* Age < 55 years
* Self-reported dialysis or renal failure
* Cognitive impairment as evaluated by study staff
* Failure to provide consent
* Failure to meet all inclusion criteria

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

SECONDARY OUTCOMES:
Proportion of participants with blood pressure within range | 10 months
Number of physician visits | 10 months
Number of emergency department visits | 10 months
Comfort with technology | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Helaine E Resnick, PhD, MPH, Principal Investigator — Association of Homes and Services for the Aging
Locations (4):
- United States (4):
  - Logan County Friendly Senior Center, Bellefontaine, Ohio
  - Miamisburg Senior Adult Center, Miamisburg, Ohio
  - Spring Valley Senior Center, Spring Valley, Ohio
  - Urbana-Champaign County Senior Center, Urbana, Ohio